CLINICAL TRIAL: NCT01289132
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Dose-Ranging Study of the Efficacy, Safety and Tolerability of TAK-536 in Subjects With Mild to Moderate Uncomplicated Essential Hypertension
Brief Title: Efficacy and Safety of Azilsartan in Participants With Mild to Moderate Uncomplicated Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. Manager, Clinical Planning, Takeda Pharmaceutical Company Limited (Japan)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-536/CCT-001; U1111-1118-3346 (Registry Identifier: WHO)
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2011-02

CONDITIONS: Essential Hypertension
Keywords: Drug Therapy
MeSH Terms: conditions — Essential Hypertension | interventions — azilsartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Azilsartan 5 mg QD (Experimental)
  Interventions: Drug: Azilsartan
- Azilsartan 10 mg QD (Experimental)
  Interventions: Drug: Azilsartan
- Azilsartan 20 mg QD (Experimental)
  Interventions: Drug: Azilsartan
- Azilsartan 40 mg QD (Experimental)
  Interventions: Drug: Azilsartan
- Azilsartan 80 mg QD (Experimental)
  Interventions: Drug: Azilsartan
- Candesartan Cilexetil 8 mg titrated to12 mg QD (Active Comparator)
  Interventions: Drug: Candesartan cilexetil

INTERVENTIONS:
Drug: Placebo — Placebo-matching tablets, orally, once daily for up to 12 weeks.
  Arms: Placebo
Drug: Azilsartan — Azilsartan 5 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: TAK-536
  Arms: Azilsartan 5 mg QD
Drug: Azilsartan — Azilsartan 10 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: TAK-536
  Arms: Azilsartan 10 mg QD
Drug: Azilsartan — Azilsartan 20 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: TAK-536
  Arms: Azilsartan 20 mg QD
Drug: Azilsartan — Azilsartan 40 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: TAK-536
  Arms: Azilsartan 40 mg QD
Drug: Azilsartan — Azilsartan 80 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: TAK-536
  Arms: Azilsartan 80 mg QD
Drug: Candesartan cilexetil — Candesartan cilexetil 8 mg, tablets, orally, once daily for 4 weeks; titrated to 12 mg, tablets, orally, once daily for up to 8 weeks.
  Other Names: Blopress®; TCV-116
  Arms: Candesartan Cilexetil 8 mg titrated to12 mg QD

SUMMARY:
The purpose of this study was to evaluate the dose-response relationships of azilsartan, once daily (QD) in participants with mild to moderate uncomplicated essential hypertension.

DETAILED DESCRIPTION:
Hypertension is known to cause multiple organ damage by being combined with not only blood pressure but also other hemodynamics, endocrinological/metabolic abnormalities and genetic factors. This becomes a medically and medical-economically significant problem in Japan The significance of early treatment of hypertension and of long-term control of blood pressure has been increasing year by year.

Takeda Pharmaceutical Company Limited invented TAK-536 (azilsartan), an angiotensin II receptor blocker for decreasing blood pressure. This study investigating the efficacy and safety of azilsartan using candesartan cilexetil, a widely used antihypertensive drug, as a reference control.

ELIGIBILITY:
Inclusion Criteria:

* Has mild to moderate uncomplicated essential hypertension.
* Has a sitting diastolic blood pressure between 95 and <110 mmHg and sitting systolic blood pressure between 150 and <180 mmHg at placebo run-in period (Week -2) or randomization visit.

Exclusion Criteria:

* Has a cardiovascular disease or symptoms
* Has been treated with more than 3 different antihypertensives within 27 days prior to placebo run-in period.
* Has a significant hepatic disorder, hyperkalemia, malignant tumor or significant renal impairment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 926 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Sitting Trough Diastolic Blood Pressure (Week 12). | Baseline and Week 12.
  The change between sitting trough clinic diastolic blood pressure measured at week 12 or final visit from diastolic blood pressure measured at baseline. Trough is a time point immediately before the next administration where drug blood concentration is lowest. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.

SECONDARY OUTCOMES:
Change from Baseline in Sitting Trough Diastolic Blood Pressure (Week 2). | Baseline and Week 2.
  The change between sitting trough clinic diastolic blood pressure measured at week 2 from diastolic blood pressure measured at baseline. Trough is a time point immediately before the next administration where drug blood concentration is lowest. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.
Change from Baseline in Sitting Trough Diastolic Blood Pressure (Week 4). | Baseline and Week 4.
  The change between sitting trough clinic diastolic blood pressure measured at week 4 from diastolic blood pressure measured at baseline. Trough is a time point immediately before the next administration where drug blood concentration is lowest. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.
Change from Baseline in Sitting Trough Diastolic Blood Pressure (Week 6). | Baseline and Week 6.
  The change between sitting trough clinic diastolic blood pressure measured at week 6 from diastolic blood pressure measured at baseline. Trough is a time point immediately before the next administration where drug blood concentration is lowest. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.
Change from Baseline in Sitting Trough Diastolic Blood Pressure (Week 8). | Baseline and Week 8.
  The change between sitting trough clinic diastolic blood pressure measured at week 8 from diastolic blood pressure measured at baseline. Trough is a time point immediately before the next administration where drug blood concentration is lowest. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.
Change from Baseline in Sitting Trough Diastolic Blood Pressure (Week 10). | Baseline and Week 10.
  The change between sitting trough clinic diastolic blood pressure measured at week 10 from diastolic blood pressure measured at baseline. Trough is a time point immediately before the next administration where drug blood concentration is lowest. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.
Change from Baseline in Sitting Trough Systolic Blood Pressure (Week 2). | Baseline and Week 2.
  The change between sitting trough clinic systolic blood pressure measured at week 2 from systolic blood pressure measured at baseline. Trough is a time point immediately before the next administration where drug blood concentration is lowest. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.
Change from Baseline in Sitting Trough Systolic Blood Pressure (Week 4). | Baseline and Week 4.
  The change between sitting trough clinic systolic blood pressure measured at week 4 from systolic blood pressure measured at baseline. Trough is a time point immediately before the next administration where drug blood concentration is lowest. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.
Change from Baseline in Sitting Trough Systolic Blood Pressure (Week 6). | Baseline and Week 6.
  The change between sitting trough clinic systolic blood pressure measured at week 6 from systolic blood pressure measured at baseline. Trough is a time point immediately before the next administration where drug blood concentration is lowest. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.
Change from Baseline in Sitting Trough Systolic Blood Pressure (Week 8). | Baseline and Week 8.
  The change between sitting trough clinic systolic blood pressure measured at week 8 from systolic blood pressure measured at baseline. Trough is a time point immediately before the next administration where drug blood concentration is lowest. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.
Change from Baseline in Sitting Trough Systolic Blood Pressure (Week 10). | Baseline and Week 10.
  The change between sitting trough clinic systolic blood pressure measured at week 10 from systolic blood pressure measured at baseline. Trough is a time point immediately before the next administration where drug blood concentration is lowest. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.
Change from Baseline in Sitting Trough Systolic Blood Pressure (Week 12). | Baseline and Week 12.
  The change between sitting trough clinic systolic blood pressure measured at week 12 or final visit from systolic blood pressure measured at baseline. Trough is a time point immediately before the next administration where drug blood concentration is lowest. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.
Number of Participants with a ≥20 mmHg Decrease in Sitting Trough Systolic Blood Pressure and a ≥10 mmHg Decrease in Sitting Trough Diastolic Blood Pressure. | Baseline and Week 12.
  Number of participants designated as responders who have a ≥20 mmHg Decrease in sitting trough systolic blood pressure and a ≥10 mmHg Decrease in sitting trough diastolic blood pressure at week 12 or final visit from baseline.
Number of Participants with a Sitting Trough Systolic Blood Pressure of <130 mmHg and a Sitting Trough Diastolic Blood Pressure of <85 mmHg. | Baseline and Week 12.
  Number of participants designated as responders with a sitting trough systolic blood pressure of <130 mmHg and a sitting trough diastolic blood pressure of <85 mmHg at week 12 or final visit from baseline.
Incidence of Adverse Events. | On occurrence (up to Week 12).
  Treatment-emergent adverse events (TEAE) are adverse events with an onset that occurs after receiving study drug and within 30 days after receiving the last dose of study drug. A TEAE may also be a pretreatment adverse event or a concurrent medical condition diagnosed prior to the date of first dose of study drug that increases in severity after the start of dosing.
Change from Baseline in Supine Systolic Blood Pressure. | Baseline and Week 12.
  The change between supine systolic blood pressure measured at week 12 or final visit from baseline. Supine systolic blood pressure is measured in participants laying on their back in a face-up position once after resting for 2 minutes.
Change from Baseline in Supine Diastolic Blood Pressure. | Baseline and Week 12.
  The change between supine diastolic blood pressure measured at week 12 or final visit from baseline. Supine diastolic blood pressure is measured in participants laying on their back in a face-up position once after resting for 2 minutes.
Change from Baseline in Standing Systolic Blood Pressure. | Baseline and Week 12.
  The change between standing systolic blood pressure measured at week 12 or final visit from baseline. Standing systolic blood pressure is measured once after participants keep a standing position for 1 minute.
Change from Baseline in Standing Diastolic Blood Pressure. | Baseline and Week 12.
  The change between standing diastolic blood pressure measured at week 12 or final visit from baseline. Standing diastolic blood pressure is measured once after participants keep a standing position for 1 minute.
Change from Baseline in Sitting Pulse Rate. | Baseline and Week 12.
  The change between sitting pulse rate measured at week 12 or final visit from baseline. Sitting pulse rate is measured at least 3 times in 1- to 2-minute intervals after sitting ≥5 minutes, repeated until 2 consecutive stable measurements are obtained.
Change from Baseline in Weight. | Baseline and Week 12.
  The change between weight recorded at week 12 or final visit from baseline.
Change from Baseline in Resting 12-lead Electrocardiogram. | Baseline and Week 12.
  The change between electrocardiogram recorded at week 12 or final visit from baseline. Electrocardiogram interpreted using one of the following categories: within normal limits, abnormal but not clinically significant, or abnormal and clinically significant.
Number of Participants with a Markedly Abnormal Blood Urea Nitrogen Clinical Laboratory Value. | Baseline and Week 12.
  The number of participants with a markedly abnormal blood urea value nitrogen collected at week 12 or final visit from baseline.
Number of Participants with a Markedly Abnormal Uric Acid Clinical Laboratory Value. | Baseline and Week 12.
  The number of participants with a markedly abnormal uric acid value collected at week 12 or final visit from baseline.
Number of Participants with a Markedly Abnormal Creatinine Clinical Laboratory Value. | Baseline and Week 12.
  The number of participants with a markedly abnormal creatinine value collected at week 12 or final visit from baseline.
Number of Participants with a Markedly Abnormal Creatine Kinase Clinical Laboratory Value. | Baseline and Week 12.
  The number of participants with a markedly abnormal creatine kinase value collected at week 12 or final visit from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Geriatric Medicine and Nephrology, Study Director — Osaka University Graduate School of Medicine